CLINICAL TRIAL: NCT05971355
Title: Clinical Comparison of LimpiAD Cream 2.5% Plus, Vehicle and an Emollient in Pediatric Patients With Atopic Dermatitis
Brief Title: Comparison of LimpiAD Cream 2.5% Plus Versus Vehicle and an Emollient in Patients With Atopic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aileens Pharma SRL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAD-09-20
Record Dates: First submitted 2021-04-27; First posted 2023-08-02 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; topical treatment; pediatric atopic dermatitis; atopic eczema; LimpiAD
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Emollients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group (Experimental): LimpiAD cream 2,5% plus to be applied twice a day (morning and evening) for 4 weeks.
  Interventions: Device: LimpiAD cream 2,5% plus
- Control group (Active Comparator): Vehicle of LimpiAD cream 2,5% plus to be applied twice a day (morning and evening) for 4 weeks.
  Interventions: Other: Vehicle
- Emollient group (Active Comparator): Emollient cream to be applied twice a day (morning and evening) for 4 weeks.
  Interventions: Other: Emollient

INTERVENTIONS:
Device: LimpiAD cream 2,5% plus — A topical formulation that contains Hyaluronic Acid conjugated with a bacterial wall fragment of Cutibacterium species (HAc-40) and an emollient base. LimpiAD exerts its post-biotic action through the seizure/ trapping and inactivation of catabolites and / or toxins produced by S. aureus as well as protecting the hydrolipidic film, especially in case of dryness, itching, and, in conditions of altered microbiome
  Arms: Treatment group
Other: Vehicle — Vehicle of LimpiAD cream 2.5 % plus which has the qualities of an emollient technically enriched with active ingredients known for their use in AD ("plus" emollient) - having the same ingredients of LimpiAD 2.5% Plus cream but without the HAc-40 component.
  Arms: Control group
Other: Emollient — Standard emollient used as neutral control, having only a moisturizing and skin barrier action, which represents the basic standard treatment (basic therapy) of atopic dermatitis according to the European Guidelines.
  Arms: Emollient group

SUMMARY:
The purpose of this randomized clinical trial is to assess the efficacy and tolerability of LimpiAD, a medical device in the form of a 2.5% Plus cream, as compared to the Vehicle of LimpiAD 2.5% Plus cream and a standard emollient used as neutral control, which represents the basic standard treatment (basic therapy) of AD according to European Guidelines in pediatric subjects with mild to moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to assess the efficacy and tolerability of LimpiAD, a medical device in the form of a 2.5% Plus cream, as compared to the Vehicle of LimpiAD 2.5% Plus cream and a standard emollient used as neutral control, which represents the basic standard treatment (basic therapy) of AD according to European Guidelines in pediatric subjects with mild to moderate Atopic Dermatitis.

This is a randomized, double-blind, multicenter, stratified, clinical trial of the medical device LimpiAD 2.5% Plus cream versus the vehicle of this medical device and versus an emollient in pedriatic Atopic Dermatitis patients that will be randomized in a 2:2:1 fashion to the compound mentioned above.

The study aims to enrol two hundred (200) pediatric subjects of both sexes, with an age ranging between 2 years old and 16 years old with atopic dermatitis of which at least 50 with mild severity (EASI 1.0-7.0 and IGA = 2) and 50 cases with moderate severity (EASI 7.1-21.0 and IGA = 3).

The treatment with the study product or with the control products shall be performed twice daily (morning and evening) after cleansing, for 4 weeks.

Clinical assessments shall be performed at baseline (T0) and after 2 and 4 weeks (T2 and T4) by means of a daily reminder diary.

The primary endpoint is the EASI improvement. The improvement shall be calculated by comparing the baseline value (T0) with the corresponding value at week 4 (T4) for LimpiAD 2.5% Plus cream versus the vehicle of LimpiAD 2.5% Plus cream and versus the emollient, in terms of detected score reduction (total EASI score).

ELIGIBILITY:
Inclusion criteria

Subjects of both sexes, with age ranging between 2 years and 16 years, Caucasian and in good health, whose parents/tutors provided a written and signed informed consent for their participation in the study shall be enrolled. In particular, as regards parents/tutors:

* both parents/tutors, in case of joint custody, should provide a written and signed informed consent for the participation of the child in the study, according to the instructions provided by the Investigators.
* they should accept to bring the child to the clinical trial facility on predefined visit days, according to the instructions provided by the Investigators;
* they should be willing and able to follow the trial requirements provided by the Investigators.

Inclusion criteria provide that:

* Symptoms and signs compatible with a clinical diagnosis of Atopic Dermatitis should be present upon enrollment;
* The clinical severity of AD should correspond to an EASI ranging between 1.0 and 21.0 and an IGA equal to 2 or 3;
* Pruritus severity assessed by means of VAS scale ≥ 4 cm) should be referred to the part of the body to be treated, as a requirement for inclusion in the study;
* The clinical assessment should envisage for the patient the indication of a moisturizing/emollient treatment as single therapy for AD (in accordance with European Guidelines on AD treatment).

Exclusion Criteria

The following items are to be considered as exclusion criteria:

* the application of cortisone-based products on the skin to be treated in the 2 weeks prior to treatment;
* use of antibiotics and systemic anti-inflammatory drugs for AD in the 2 weeks preceding treatment and during the study (paracetamol is allowed at dosages and indications recommended for use as an antipyretic and analgesic);
* ongoing baseline treatment (T0) with anti-inflammatory drugs, antihistamines, antitussives and/or inhaled steroids in the 2 previous weeks, retinoids and/or immunosuppressants in the previous 6 months.
* use of systemic steroids in the 4 weeks prior to the study.
* Intense and prolonged sun exposure in the 30 days preceding the screening.
* severe AD (EASI > 21) or mild/moderate AD requiring a local and/or systemic treatment included among treatments not allowed, as provided for in exclusion criteria;
* hypersensitivity to the study products.
* acute or chronic skin diseases - except for atopic eczema - which may invalidate clinical assessments or overlap with AD skin picture;
* systemic diseases which may affect the subject's safety or wellbeing or interfere with skin response.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  The change shall be calculated by comparing the baseline value (T0) with the corresponding value at 4 weeks (T4) for LimpiAD cream 2,5% Plus versus the Vehicle of LimpiAD cream 2,5% Plus in terms of detected score reduction (total EASI score).
  INTERPRET EASI: Clear 0; Almost clear 0.1-1.0 ; Mild 1.1-7.0 ; Moderate 7.1-21.0 ; Severe 21.1-50.0; Very severe 50.1-72.0

SECONDARY OUTCOMES:
Change in Investigator Global Assessment (IGA) scale for Atopic Dermatitis | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  The change shall be calculated by comparing the baseline value (T0) with the corresponding values at 2 weeks (T2) and 4 weeks (T4) in the treatment arm with LimpiAD cream 2.5% Plus as compared to the other 2 study treatment arms.
  INTERPRET IGA: 0 - Not affected; 1 - Little affected; 2 - Mild erythema; 3 - Moderate erythema; 4 - Severe Marked erythema
Eczema Area and Severity Index (EASI) Change | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  The change shall be calculated, by comparing the baseline value (T0) with the corresponding values at 2 weeks (T2) and 4 weeks (T4) in the treatment arm with LimpiAD cream 2.5% Plus as compared to the other 2 study treatment arms in terms of:
  - % of patients reaching a 50% (EASI50), 75% (EASI75), 90% (EASI90) and 100% (EASI100) reduction in the baseline score.
  INTERPRET EASI: Clear 0; Almost clear 0.1-1.0 ; Mild 1.1-7.0 ; Moderate 7.1-21.0 ; Severe 21.1-50.0; Very severe 50.1-72.0
Change in pruritus at the 4 week (T4) | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  Change in pruritus at the 4th week (T4): by improvement we mean a Visual Analogue Scale (VAS) reduction below 4 cm, with at least 2-score deviation from baseline (T0), including only the cases with VAS > 5 at baseline, in the treatment arm with LimpiAD cream 2.5% Plus as compared to the other 2 study treatment arms.
  In the visual analogue scale (VAS), patients are asked to mark on a 10-cm ruler ranging from 0 (no itch) to 10 (worst imaginable itch).
Change in sleep at 4 weeks (T4) | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  Change in sleep at 4 weeks (T4) intended as mean a Visual Analogue Scale (VAS) reduction below 4 cm, with at least 2-score deviation from baseline (T0), including only the cases with VAS >5 cm at baseline, in the treatment arm with LimpiAD cream 2.5% Plus as compared to the other 2 study treatment arms.
  In the visual analogue scale (VAS), patients are asked to mark on a 10-cm ruler ranging from 0 (no disturbance sleep) to 10 (very much disturbed sleep).
Change in extension and signs intensity of the target areas | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  Change in extension and signs intensity of the target areas, assessed as local Eczema Area and Severity Index (EASI), by separately considering the skin fold area with respect to the fold-free skin area at 2 weeks (T2) and 4 weeks (T4) in the treatment arm with LimpiAD cream 2.5% Plus as compared to the other 2 study treatment arms
Children's Dermatology Life Quality Index (CDLQI) questionnaire | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  Change in Children's Dermatology Life Quality Index (CDLQI). The change shall be calculated, by comparing the baseline total points (T0) with the corresponding total points at 2 weeks (T2) and 4 weeks (T4) in the treatment arm with LimpiAD cream 2.5% Plus as compared to the other 2 study treatment arms in terms of:
  * % of achievement of CDLQI <10
  * CDLQI average score reduction
  The CDLQI has 11 questions asking about the impact of a atopic dermatitis on the life of the affected child over the last week.
  Interpretation of QoL: 0-2 = no effect on QoL, 3-7 small effect, 8-13 moderate effect, 14-19 very large effect, 20-33 extremely large effect
Microbial balance | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  Change in Cutibacterium acne/Staphylococcus ratio on the affected skin in the treatment arm with LimpiAD cream 2.5% Plus as compared to the other 2 study treatment arms.
Functional recovery | Baseline (T0), 2 weeks (T2) and 4 weeks (T4)
  Functional recovery:
  - change in vascularization measured by dynamic OCT (D-OCT) imaging, assessed in a subsample of subjects, in the treatment arm with LimpiAD 2.5% cream Plus as compared to the other 2 study treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Farnetani, Prof, Principal Investigator — University of Modena e Reggio Emilia
Locations (5):
- Italy (5):
  - University of Bari Hospital, Bari
  - University of Modena e Reggio Emilia, Modena
  - University of Naples Hospital, Naples
  - S. Gallicano Hospital, Rome
  - University Rome La Sapienza (Hospital Umberto I), Rome

IPD SHARING:
Plan to Share IPD: No